CLINICAL TRIAL: NCT00190749
Title: Insulin Sensitivity in Patients With Schizophrenia or Schizoaffective Disorder Treated With Olanzapine and Risperidone
Brief Title: Safety Study of Olanzapine and a Comparator in Patients With Schizophrenia and Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5296; F1D-MC-S014 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-07-23 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine (Experimental)
  Interventions: Drug: olanzapine
- Risperidone (Active Comparator)
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: olanzapine — 5-20 mg, oral, capsules, daily, 12 weeks.
  Other Names: LY170053; Zyprexa
  Arms: Olanzapine
Drug: risperidone — 2-6 mg, oral, capsules, twice daily (BID), 12 weeks.
  Arms: Risperidone

SUMMARY:
This study will assess whether olanzapine and/or risperidone affect the way the human body uses sugar in the blood.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Diagnosed with Schizophrenia or Schizoaffective disorder
* Ability to visit the doctor's office for scheduled visits

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Have a body mass index (BMI) greater than 40
* Have diabetes, heart disease or any other unstable illness
* Have known positive human immunodeficiency virus (HIV)
* Are currently taking olanzapine, risperidone, clozapine, glucocorticoids, injectable antipsychotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2003-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California, United States

REFERENCES:
- [Derived] Case M, Treuer T, Karagianis J, Hoffmann VP. The potential role of appetite in predicting weight changes during treatment with olanzapine. BMC Psychiatry. 2010 Sep 14;10:72. doi: 10.1186/1471-244X-10-72. PMID 20840778
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period I was a Screening Period. Study Period II was a Inpatient Washout/Diet Stabilization Period. Study Period III (randomization) was the Double-Blind Therapy Period.
Groups:
- Olanzapine: Olanzapine, 5-20 mg, oral, capsules, daily, 12 weeks.
- Risperidone: Risperidone, 2-6 mg, oral, capsules, twice daily (BID), 12 weeks.
Period: Overall Study
Arm/Group | Olanzapine | Risperidone
Started | 68 | 62
Completed | 42 | 31
Not Completed | 26 | 31
Not completed — Lost to Follow-up | 8 | 11
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Protocol Violation | 5 | 4
Not completed — Adverse Event | 0 | 5
Not completed — Lack of Efficacy | 2 | 3
Not completed — Reason Not Specified | 0 | 2
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Risperidone | Total
Number analyzed (Participants) | 68 | 62 | 130
Age Continuous [Mean (Standard Deviation); unit: years] | 43.49 (9.45) | 42.58 (8.98) | 43.06 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 45 | 41 | 86
Region of Enrollment [Number; unit: participants]
  United States | 68 | 62 | 130
Diagnosis [Number; unit: participants]
  Schizophrenia,paranoid | 40 | 45 | 85
  Schizoaffective disorder | 27 | 16 | 43
  Schizophrenia, undifferentiated | 1 | 1 | 2
Race/Ethnicity [Number; unit: participants]
  Caucasian | 27 | 30 | 57
  African descent | 34 | 26 | 60
  Hispanic | 4 | 5 | 9
  East Asian | 1 | 0 | 1
  Other | 2 | 1 | 3
Brief Psychiatric Rating Scale Anxiety Depression Score-Baseline [Mean (Standard Deviation); unit: units on a scale] — Brief Psychiatric Rating Scale (BPRS) Anxiety-Depression Score assesses the degree of severity of a subject's anxiety-depression symptoms. BPRS Anxiety-Depression Score is the sum of Item Scores 1, 2, 5 and 9. Item scores range from 0 (not present) to 6 (extremely severe). Total Scores for Anxiety-Depression range from 0 to 24.
  units on a scale | 4.46 (2.46) | 3.74 (2.13) | 4.12 (2.33)
Brief Psychiatric Rating Scale Negative Symptom Score-Baseline [Mean (Standard Deviation); unit: units on a scale] — Brief Psychiatric Rating Scale (BPRS) Negative Score assesses the degree of severity of a subject's negative symptoms. BPRS Negative Score is the sum of Item Scores 3, 13, and 16. Item scores range from 0 (not present) to 6 (extremely severe). Total Scores for Negative Score range from 0 to 18.
  units on a scale | 2.28 (1.98) | 1.89 (1.79) | 2.09 (1.89)
Brief Psychiatric Rating Scale Positive Symptom Score-Baseline [Mean (Standard Deviation); unit: units on a scale] — Brief Psychiatric Rating Scale (BPRS) Positive Score assesses the degree of severity of a subject's positive symptoms. BPRS Positive Score is the sum of Item Scores 4, 11, 12, and 15. Item scores range from 0 (not present) to 6 (extremely severe). Total Scores for Positive Score range from 0 to 24.
  units on a scale | 5.40 (2.69) | 5.47 (2.52) | 5.43 (2.60)
Brief Psychiatric Rating Scale Total Score-Baseline [Mean (Standard Deviation); unit: units on a scale] — Brief Psychiatric Rating Scale (BPRS) Total Score is an 18-item clinician-administered scale used to assess the degree of severity of a subject's general psychopathological symptoms. Item scores range from 0 (not present) to 6 (extremely severe). Total Scores range from 0 to 108.
  units on a scale | 15.63 (6.06) | 14.29 (6.00) | 14.99 (6.04)
Clinical Global Impression Severity Score- Baseline [Mean (Standard Deviation); unit: units on a scale] — Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 3.68 (0.56) | 3.65 (0.52) | 3.66 (0.54)
Extrapyramidal Scores/Abnormal Involuntary Movement-Baseline [Mean (Standard Deviation); unit: units on a scale] — A 12-item instrument assesses observed abnormal movements in different parts of body. Seven items are scored in a 5-point scale (0 = none/normal, 4 = severe) which evaluates abnormal movements in 3 main anatomic areas (orofacial area, extremities, and trunk). Total scores range from 0 to 28. Five collected elements are not used in this total.
  units on a scale | 0.42 (1.14) | 0.47 (1.13) | 0.44 (1.13)
Extrapyramidal Scores/Barnes Akathisia Rating Scale (BARS) Global Clinical Assessment-Baseline [Mean (Standard Deviation); unit: units on a scale] — The BARS is a 4-item instrument that evaluates akathisia associated with use of antipsychotic medications. Item 4 is the Global clinical assessment and is rated 0 to 5 (0 = absent, 5 = severe).
  units on a scale | 0.27 (0.66) | 0.32 (0.67) | 0.29 (0.67)
Extrapyramidal Scores/Simpson-Angus-Baseline [Mean (Standard Deviation); unit: units on a scale] — Measures neuroleptic-induced parkinsonism. Total score of Simpson Angus Scale consists of the sum of 10 itemsrated on a 5-point severity scale where 0=normal and 4=extreme. The total score ranges from 0 to 40.
  units on a scale | 0.97 (1.87) | 0.90 (1.80) | 0.94 (1.83)

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline to Last Observation In Normalized Insulin Sensitivity Index at Low Insulin Phase Using Change in Weight as a Covariate
Description: Normalized insulin sensitivity index (Mffm/I) was defined as the ratio of whole body glucose disposal rate normalized to fat-free mass (Mffm) divided by the plasma insulin concentration (I) during steady-state conditions of the clamp procedure. Units:[(mg glucose)*min*mL] / [(kg fat free body mass)*(micro IU insulin)]
Time Frame: baseline and 12 weeks
Population: N=number of patients with a baseline and post-baseline result within each treatment group for Mffm/I and weight.
Measure: Mean (Standard Deviation); unit: Mffm/I
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 41 | 33
Mffm/I
  Baseline | 0.1664 (0.1120) | 0.1937 (0.1286)
  Change to Last Observation | -0.0149 (0.0786) | -0.0327 (0.0829)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.226, t-test, 2 sided — P-value for change to last observation
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.030, t-test, 2 sided — P-value is change to last observation
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.204, ANCOVA — P-value for change to last observation

2. Secondary Outcome: Pairwise Correlations Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in Weight.
Description: Normalized insulin sensitivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in Mffm/I and changes in weight
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 41 | 33
correlation | -0.212 | -0.188
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.184, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.295, Pearson's correlation coefficient

3. Secondary Outcome: Pairwise Correlations Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in Body Mass Index (BMI)
Description: Normalized insulin sensitivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in Mffm/I and changes in BMI
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 41 | 33
correlation | -0.182 | -0.195
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.256, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.277, Pearson's correlation coefficient

4. Secondary Outcome: Pairwise Correlations Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in Ratio of Visceral Fat Area to the Subcutaneous Fat Area.
Description: Normalized insulin sensitivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in ratio of visceral far area to subcutaneous fat area
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 32 | 26
correlation | -0.055 | 0.101
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.766, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.622, Pearson's correlation coefficient

5. Secondary Outcome: Pairwise Correlations Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in Brief Psychiatric Rating Scale Scores.
Description: Normalized insulin senstivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in Mffm/I and changes in Brief Psychiatric Rating Scale scores
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 41 | 33
correlation | 0.035 | 0.066
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.829, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.714, Pearson's correlation coefficient

6. Secondary Outcome: Pairwise Correlations Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in Clinical Global Impression - Severity of Illness Scale Scores.
Description: Normalized insulin sensitivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in Mffm/I and changes in Clinical Global Impression-Severity of Illness scale scores
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 41 | 33
correlation | 0.068 | 0.234
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.672, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.191, Pearson's correlation coefficient

7. Secondary Outcome: Pairwise Correlations Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in Abnormal Involuntary Movement Scale Scores.
Description: Normalized insulin sensitivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in Mffm/I and changes in Abnormal Involuntary Movement Scale scores
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 41 | 33
correlation | 0.001 | -0.134
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.994, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.456, Pearson's correlation coefficient

8. Secondary Outcome: Pairwise Correlation Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in Barnes Akathisia Scale Scores.
Description: Normalized insulin sensitivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in Mffm/I and changes in Barnes Akathisia scores
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 41 | 33
correlation | -0.120 | 0.006
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.454, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.974, Pearson's correlation coefficient

9. Secondary Outcome: Pairwise Correlations Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in the Simpson Angus Scale Scores.
Description: Normalized insulin sensitivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in the Simpson Angus Scale scores
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 41 | 33
correlation | 0.184 | 0.249
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.249, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.163, Pearson's correlation coefficient

10. Secondary Outcome: Pairwise Correlations Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in Waist Circumference.
Description: Normalized insulin sensitivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in Mffm/I and changes in waist circumference
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 40 | 29
correlation | -0.206 | -0.263
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.201, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.168, Pearson's correlation coefficient

11. Secondary Outcome: Pairwise Correlations Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in Visceral Fat Area.
Description: Normalized insulin sensitivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in Mffm/I and changes in visceral fat area
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 32 | 27
correlation | -0.048 | -0.057
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.793, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.777, Pearson's correlation coefficient

12. Secondary Outcome: Pairwise Correlations Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in Subcutaneous Fat Area.
Description: Normalized insulin sensitivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in Mffm/I and changes in subcutaneous fat area
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 32 | 27
correlation | -0.043 | -0.085
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.815, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.675, Pearson's correlation coefficient

13. Secondary Outcome: Pairwise Correlations Between Between Changes in Normalized Insulin Sensitivity Index at Low Insulin Phase and Changes in Eating Behavior Assessment Scale Scores.
Description: Normalized insulin sensitivity index (Mffm/I) at low insulin phase-pairwise correlations between changes in Mffm/I and changes in Eating Behavior Assessment Scale scores
Time Frame: 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Number; unit: correlation
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 41 | 33
correlation
  Item 1: How Hungry? | -0.137 | -0.371
  Item 2: How Strong Appetite? | -0.137 | -0.269
  Item 3: Craved Sweets or Other Carbohydrates? | -0.009 | 0.035
  Item 4: Craved Fatty Foods? | -0.068 | -0.184
  Item 5: Felt Full or Satisfied After Meal? | -0.117 | -0.060
  Item 6:Excessive Amount of Food to Feel Satisfied? | 0.134 | 0.067
  Item 7: Thinking About Food? | -0.172 | 0.045
  Item 8: Overeating? | -0.032 | -0.165
  Item 9: Feel Eating is Out of Control? | -0.075 | -0.354
Statistical Analysis 1: Comparison: Olanzapine; Change in Eating Behavior Item 1; Test type: Superiority or Other; p = 0.393, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Risperidone; Change in Eating Behavior Item 1; Test type: Superiority or Other; p = 0.033, Pearson's correlation coefficient
Statistical Analysis 3: Comparison: Olanzapine; Change in Eating Behavior Item 2; Test type: Superiority or Other; p = 0.392, Pearson's correlation coefficient
Statistical Analysis 4: Comparison: Risperidone; Change in Eating Behavior Item 2; Test type: Superiority or Other; p = 0.129, Pearson's correlation coefficient
Statistical Analysis 5: Comparison: Olanzapine; Change in Eating Bahavior Item 3; Test type: Superiority or Other; p = 0.956, Pearson's correlation coefficient
Statistical Analysis 6: Comparison: Risperidone; Change in Eating Behavior Item 3; Test type: Superiority or Other; p = 0.846, Pearson's correlation coefficient
Statistical Analysis 7: Comparison: Olanzapine; Change in Eating Behavior Item 4; Test type: Superiority or Other; p = 0.675, Pearson's correlation coefficient
Statistical Analysis 8: Comparison: Risperidone; Change in Eating Behavior Item 4; Test type: Superiority or Other; p = 0.306, Pearson's correlation coefficient
Statistical Analysis 9: Comparison: Olanzapine; Change in Eating Behavior Item 5; Test type: Superiority or Other; p = 0.468, Pearson's correlation coefficient
Statistical Analysis 10: Comparison: Risperidone; Change in Eating Behavior Item 5; Test type: Superiority or Other; p = 0.739, Pearson's correlation coefficient
Statistical Analysis 11: Comparison: Olanzapine; Change in Eating Behavior Item 6; Test type: Superiority or Other; p = 0.404, Pearson's correlation coefficient
Statistical Analysis 12: Comparison: Risperidone; Change in Eating Behavior Item 6; Test type: Superiority or Other; p = 0.711, Pearson's correlation coefficient
Statistical Analysis 13: Comparison: Olanzapine; Change in Eating Behavior Item 7; Test type: Superiority or Other; p = 0.281, Pearson's correlation coefficient
Statistical Analysis 14: Comparison: Risperidone; Change in Eating Behavior Item 7; Test type: Superiority or Other; p = 0.805, Pearson's correlation coefficient
Statistical Analysis 15: Comparison: Olanzapine; Change in Eating Behavior Item 8; Test type: Superiority or Other; p = 0.844, Pearson's correlation coefficient
Statistical Analysis 16: Comparison: Risperidone; Change in Eating Bahavior Item 8; Test type: Superiority or Other; p = 0.359, Pearson's correlation coefficient
Statistical Analysis 17: Comparison: Olanzapine; Change in Eating Behavior Item 9; Test type: Superiority or Other; p = 0.642, Pearson's correlation coefficient
Statistical Analysis 18: Comparison: Risperidone; Change in Eating Behavior Item 9; Test type: Superiority or Other; p = 0.043, Pearson's correlation coefficient

14. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Body Mass Index
Description: Within-and Between-Treatment Group changes in Body Mass Index from baseline to last observation carried forward.
Time Frame: baseline and 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations
Measure: Mean (Standard Deviation); unit: kilograms per square meter (kg/m2)
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 41 | 33
kilograms per square meter (kg/m2)
  Baseline | 28.96 (5.17) | 28.79 (5.40)
  Change to Last Observation | 1.02 (1.61) | 0.39 (1.15)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p < .001, t-test, 2 sided; Within group p-values are from t-tests on Least Squares Mean (LSMean) change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.019, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.065, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change =Baseline Treatment Pooled Investigator

15. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Weight
Description: Weight change from baseline to last visit (last observation carried forward)
Time Frame: baseline and 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 41 | 33
kilograms
  Baseline | 85.93 (17.26) | 86.55 (19.53)
  Change to Last Observation | 2.98 (4.82) | 1.23 (4.45)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p < .001, t-test, 2 sided; With group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.013, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.076, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change = Baseline Treatment Pooled Investigator

16. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Waist Circumference
Description: Waist circumference change from baseline to last observation carried forward.
Time Frame: baseline and 12 weeks
Population: Randomized patients who completed the baseline and endpoint clamps with both diet stabilizations.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 40 | 29
centimeters
  Baseline | 99.13 (14.42) | 98.49 (11.60)
  Change to Last Observation | 2.38 (7.46) | 0.17 (4.99)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.007, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.266, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.239, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change = Baseline Treatment Pooled Investigator

17. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Visceral Fat Area
Description: Visceral fat area change from baseline to last observation carried forward, all randomized patients, double-blind treatment period
Time Frame: baseline and 12 weeks
Population: Abdominal CT scan of changes from baseline to last observation of randomized patients who completed baseline and endpoint clamps with both diet stabilizations
Measure: Mean (Standard Deviation); unit: square centimeters (cm2)
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 32 | 27
square centimeters (cm2)
  Baseline | 101.46 (54.99) | 102.17 (52.61)
  Change to Last Observation | 4.70 (21.21) | 8.70 (42.39)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.274, t-test, 2 sided; Within group p-vales are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.105, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.609, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change= Baseline Treatment Pooled Investigator

18. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Subcutaneous Fat Area
Description: Subcutaneous fat area change from baseline to last observation carried forward, all randomized patients, double-blind treatment period
Time Frame: baseline and 12 weeks
Population: Abdominal CT scan change from baseline to last observation for randomized patients who completed baseline and endpoint clamps with both diet stabilizations
Measure: Mean (Standard Deviation); unit: square centimeters (cm2)
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 32 | 27
square centimeters (cm2)
  Baseline | 281.07 (158.59) | 317.16 (172.19)
  Change to last observation | 4.94 (40.36) | 35.15 (105.64)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.406, t-test, 2 sided; With group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.011, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.076, ANCOVA; Overall group p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

19. Secondary Outcome: Change From Baseline to 12 Week Endpoint in the Ratio of the Visceral Fat Area to the Subcutaneous Fat Area
Description: Ratio of the visceral fat area to the subcutaneous fat area change from baseline to last observation carried forward, all randomized patients, double-blind treatment period
Time Frame: baseline and 12 weeks
Population: Abdominal CT scan change from baseline to last observation of randomized patients who completed the baseline and endpoint clamps with both diet stabilizations
Measure: Mean (Standard Deviation); unit: ratio in square centimeters (cm2)
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 32 | 26
ratio in square centimeters (cm2)
  Baseline | 0.41 (0.25) | 0.43 (0.33)
  Change to last observation | 0.01 (0.12) | 0.00 (0.14)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.456, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.712, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.689, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change= Baseline Treatment Pooled Investigator

20. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Brief Psychiatric Rating Scale (BPRS) Scores
Description: Brief Psychiatric Rating Scale (BPRS) is an 18-item clinician-administered scale used to assess the degree of severity of a subject's general psychopathological symptoms. Item scores range from 0 (not present) to 6 (extremely severe). Total Scores range from 0 to 108; Positive Subscale Scores range from 0 to 24. Negative Subscale Scores range from 0 to 18. Anxiety-Depression Subscale Scores range from 0 to 24.
Time Frame: baseline and 12 weeks
Population: BPRS Total and Subscale Scores-Change from Baseline to Last Observation Carried Forward, all randomized patients, double-blind treatment period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 60 | 56
units on a scale
  Total Score Baseline | 13.32 (6.26) | 13.96 (6.02)
  Total Score Change to Last Observation | -1.98 (6.30) | -1.48 (7.99)
  Positive Subscale Score Baseline | 5.22 (2.75) | 5.27 (2.51)
  Positive Subscale Score Change to Last Observation | -0.82 (2.81) | -1.20 (3.08)
  Negative Subscale Score Baseline | 2.32 (2.04) | 1.88 (1.83)
  Negative Subscale Score Change to Last Observation | -0.38 (1.58) | -0.02 (1.99)
  Anxiety-Depression Baseline | 4.33 (2.59) | 3.73 (2.18)
  Anxiety-Depression Change to Last Observation | -0.78 (2.29) | -0.32 (2.50)
Statistical Analysis 1: Comparison: Olanzapine; Total Score; Test type: Superiority or Other; p = 0.111, t-test, 2 sided; Within group p-values are from t-tests on LSMean
Statistical Analysis 2: Comparison: Risperidone; Total Score; Test type: Superiority or Other; p = 0.159, t-test, 2 sided; Within group p-values are from t-tests on LSMean changes
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Total Score; Test type: Superiority or Other; p = 0.951, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change =Baseline Treatment Pooled Investigator
Statistical Analysis 4: Comparison: Olanzapine; Positive Subscale; Test type: Superiority or Other; p = 0.012, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 5: Comparison: Risperidone; Positive subscale; Test type: Superiority or Other; p = 0.002, t-test, 2 sided; With group p-values are from t-tests on LSMean
Statistical Analysis 6: Comparison: Olanzapine vs Risperidone; Positive subscale; Test type: Superiority or Other; p = 0.467, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change =Baseline Treatment Pooled Investigator
Statistical Analysis 7: Comparison: Olanzapine; Negative subscale; Test type: Superiority or Other; p = 0.365, t-test, 2 sided; With group p-values are from t-tests on LSMean change
Statistical Analysis 8: Comparison: Risperidone; Negative subscale; Test type: Superiority or Other; p = 0.846, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 9: Comparison: Olanzapine vs Risperidone; Negative subscale; Test type: Superiority or Other; p = 0.559, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 10: Comparison: Olanzapine; Anxiety-Depression subscale; Test type: Superiority or Other; p = 0.150, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 11: Comparison: Risperidone; Anxiety-Depression subscale; Test type: Superiority or Other; p = 0.612, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 12: Comparison: Olanzapine vs Risperidone; Anxiety-Depression subscale; Test type: Superiority or Other; p = 0.475, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

21. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Clinical Global Impression - Severity of Illness Scores
Description: Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients.
Time Frame: baseline and 12 weeks
Population: Change from baseline to last observation carried forward, all randomized patients, double-blind treatment period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 60 | 56
units on a scale
  Baseline | 3.65 (0.55) | 3.61 (0.53)
  Change to last observation | -0.22 (0.58) | -0.23 (0.66)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = .012, t-test, 2 sided — Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.010, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.760, ANCOVA; Overall p-values are from Type 3 sums of square ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

22. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Abnormal Involuntary Movement Scale Scores
Description: A 12-item instrument assesses observed abnormal movements in different parts of body. Seven items are scored in a 5-point scale (0 = none/normal, 4 = severe) which evaluates abnormal movements in 3 main anatomic areas (orofacial area, extremities, and trunk). Total scores range from 0 to 28. Five collected elements are not used in this total.
Time Frame: baseline and 12 weeks
Population: Change from baseline to last observation carried forward, all randomized patients, double-blind treatment period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 54 | 47
units on a scale
  Baseline | 0.48 (1.24) | 0.53 (1.25)
  Change to last observation | 0.04 (1.15) | 0.04 (1.35)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.943, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.763, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.832, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

23. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Barnes Akathisia Rating Scale (BARS) Scores
Description: The BARS is a 4-item instrument that evaluates akathisia associated with use of antipsychotic medications. Item 4 is the Global clinical assessment and is rated 0 to 5 (0 = absent, 5 = severe). The other 3 items (related to objective and subjective assessments) are not used for these analyses.
Time Frame: baseline and 12 weeks
Population: Change from baseline to last observation carried forward, all randomized patients, double-blind treatment period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 54 | 47
units on a scale
  Baseline | 0.24 (0.64) | 0.36 (0.70)
  Change to last observation | 0.02 (0.84) | -0.02 (0.82)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.623, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.853, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.591, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

24. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Simpson Angus Scale Scores
Description: Measures neuroleptic-induced parkinsonism. Total score of Simpson Angus Scale consists of the sum of 10 items rated on a 5-point severity scale where 0=normal and 4=extreme. The total score ranges from 0 to 40.
Time Frame: baseline and 12 weeks
Population: Change from baseline to last observation carried forward, all randomized patients, double-blind treatment period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 54 | 47
units on a scale
  Baseline | 1.13 (2.02) | 0.94 (1.79)
  Change to last observation | -0.06 (1.48) | 0.30 (1.92)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.302, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.922, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.479, ANCOVA; Overall group p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

25. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Eating Behavior Assessment Scale Scores
Description: Eating Behavior Assessment Scale is a 9-item self-rated tool used to evaluate appetite and eating behaviors. Item scores range from 0 (never) to 4 (always).
Time Frame: baseline and 12 weeks
Population: Change from baseline to last observation carried forward, all randomized patients, double-blind treatment period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 59 | 53
units on a scale
  Item 1 Baseline (How Hungry?) | 1.42 (1.09) | 1.32 (0.94)
  Item 1 Change to Last Observation | 0.25 (1.27) | 0.42 (1.18)
  Item 2 Baseline (How Strong Appetite?) | 1.54 (1.10) | 1.32 (1.03)
  Item 2 Change to Last Observation | 0.17 (1.26) | 0.38 (1.33)
  Item 3 Baseline (Craved Sweets or Other Carbos?) | 1.00 (1.17) | 0.83 (1.10)
  Item 3 Change to Last Observation | 0.19 (1.47) | 0.36 (1.18)
  Item 4 Baseline (Craved Fatty Foods?) | 0.80 (1.01) | 0.74 (1.00)
  Item 4 Change to Last Observation | 0.31 (1.52) | 0.25 (1.05)
  Item 5 Baseline (Felt Full After Meal?) | 2.59 (0.93) | 2.55 (0.89)
  Item 5 Change to Last Observation | -0.17 (1.15) | 0.00 (1.19)
  Item 6 Baseline(Excessive Food to Feel Satisfied?) | 0.86 (1.21) | 0.79 (1.12)
  Item 6 Change to Last Observation | 0.17 (1.40) | 0.28 (1.25)
  Item 7 Baseline (Thinking About Food?) | 0.90 (1.18) | 0.77 (1.14)
  Item 7 Change to Last Observation | 0.12 (1.31) | 0.13 (1.36)
  Item 8 Baseline (Overeating?) | 0.42 (0.95) | 0.53 (1.08)
  Item 8 Change to Last Observation | 0.17 (1.33) | 0.15 (1.31)
  Item 9 Baseline (Feel Eating is Out of Control?) | 0.10 (0.36) | 0.26 (0.76)
  Item 9 Change to Last Observation | 0.25 (0.94) | 0.11 (1.01)
Statistical Analysis 1: Comparison: Olanzapine; Item 1; Test type: Superiority or Other; p = 0.004, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Item 1; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Item 1; Test type: Superiority or Other; p = 0.549, ANCOVA; Overall p-values are from Type 3 sums of squares, ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 4: Comparison: Olanzapine; Item 2; Test type: Superiority or Other; p = 0.011, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 5: Comparison: Risperidone; Item 2; Test type: Superiority or Other; p = 0.009, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 6: Comparison: Olanzapine vs Risperidone; Item 2; Test type: Superiority or Other; p = 0.793, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 7: Comparison: Olanzapine; Item 3; Test type: Superiority or Other; p = 0.045, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 8: Comparison: Risperidone; Item 3; Test type: Superiority or Other; p = 0.027, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 9: Comparison: Olanzapine vs Risperidone; Item 3; Test type: Superiority or Other; p = 0.699, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 10: Comparison: Olanzapine; Item 4; Test type: Superiority or Other; p = 0.002, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 11: Comparison: Risperidone; ITem 4; Test type: Superiority or Other; p = 0.019, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 12: Comparison: Olanzapine vs Risperidone; Item 4; Test type: Superiority or Other; p = 0.733, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 13: Comparison: Olanzapine; Item 5; Test type: Superiority or Other; p = 0.034, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 14: Comparison: Risperidone; Item 5; Test type: Superiority or Other; p = 0.235, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 15: Comparison: Olanzapine vs Risperidone; Item 5; Test type: Superiority or Other; p = 0.532, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 16: Comparison: Olanzapine; Item 6; Test type: Superiority or Other; p = 0.242, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 17: Comparison: Risperidone; Item 6; Test type: Superiority or Other; p = 0.186, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 18: Comparison: Olanzapine vs Risperidone; Item 6; Test type: Superiority or Other; p = 0.799, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 19: Comparison: Olanzapine; Item 7; Test type: Superiority or Other; p = 0.097, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 20: Comparison: Risperidone; Item 7; Test type: Superiority or Other; p = 0.214, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 21: Comparison: Olanzapine vs Risperidone; Item 7; Test type: Superiority or Other; p = 0.827, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 22: Comparison: Olanzapine; Item 8; Test type: Superiority or Other; p = 0.151, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 23: Comparison: Risperidone; Item 8; Test type: Superiority or Other; p = 0.071, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 24: Comparison: Olanzapine vs Risperidone; Item 8; Test type: Superiority or Other; p = 0.629, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 25: Comparison: Olanzapine; Item 9; Test type: Superiority or Other; p = 0.036, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 26: Comparison: Risperidone; Item 9; Test type: Superiority or Other; p = 0.112, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 27: Comparison: Olanzapine vs Risperidone; Item 9; Test type: Superiority or Other; p = 0.806, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

26. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Fasting Lipid Parameters Including Total Cholesterol
Description: Fasting lipid parameters including total cholesterol, change from baseline to last observation carried forward.
Time Frame: baseline and 12 weeks
Population: Change from baseline to last observation, all randomized patients, double-blind treatment period
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 51 | 49
millimoles per Liter (mmol/L)
  Baseline | 4.91 (1.06) | 4.97 (1.12)
  Change to Last Observation | 0.18 (0.89) | 0.01 (0.79)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.156, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.829, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.352, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

27. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Fasting Lipid Parameters Including Direct Low Density Lipoprotein (LDL)
Description: Fasting lipid parameters including Direct LDL, change from baseline to last observation carried forward.
Time Frame: baseline and 12 weeks
Population: Change from baseline to last observation, all randomized patients, double-blind treatment period
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 51 | 49
millimoles per Liter (mmol/L)
  Baseline | 3.18 (0.90) | 3.11 (0.99)
  Change to last observation | -0.03 (0.67) | -0.02 (0.63)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.740, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.760, t-test, 2 sided; Within group p-values are frm t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.997, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

28. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Fasting Lipid Parameters Including High Density Lipoprotein (HDL)
Description: Fasting lipid parameters including HDL change from baseline to last observation carried forward.
Time Frame: baseline and 12 weeks
Population: Change from baseline to last observation, all randomized patients, double-blind treatment period
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 51 | 48
millimoles per Liter (mmol/L)
  Baseline | 1.08 (0.25) | 1.18 (0.32)
  Change to last observation | 0.06 (0.24) | 0.05 (0.27)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.176, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.237, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.996, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

29. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Fasting Lipid Parameters Including Triglycerides
Description: Changes in fasting lipid parameters including triglycerides last observation carried forward (LOCF) mean change from baseline
Time Frame: baseline and 12 weeks
Population: Change from baseline to last observation, all randomized patients, double-blind treatment period
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 51 | 49
millimoles per Liter (mmol/L)
  Baseline | 1.68 (0.91) | 1.55 (0.85)
  Change to Last Observation | 0.34 (1.12) | -0.10 (0.74)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Superiority or Other; p = 0.027, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.545, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; Test type: Superiority or Other; p = 0.024, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

30. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Fasting Lipid Parameters Including Lipoprotein Subclasses
Description: Changes in lipid parameters and subclass lipoproteins last observation carried forward (LOCF) mean change from baseline. HDL=High Density Lipoprotein, IDL=Intermdiate Density Lipoprotein, LDL=Low Density Lipoprotein, VLDL=Very Low Density Lipoprotein.
Time Frame: baseline and 12 weeks.
Population: Mean change from baseline, all randomized patients, double-blind treatment period
Measure: Mean (Standard Deviation); unit: nanomoles per Liter (nmol/L)
Arm/Group | Olanzapine | Risperidone
Number analyzed (Participants) | 40 | 32
nanomoles per Liter (nmol/L)
  HDL particles, total, baseline | 28.39 (5.38) | 29.81 (5.29)
  HDL particles, total, change to last observation | 1.71 (4.84) | -1.09 (4.34)
  IDL, baseline | 53.18 (55.32) | 52.56 (61.38)
  IDL, change to last observation | 21.40 (59.63) | -2.69 (46.07)
  Medium small LDL, baseline | 175.15 (98.59) | 197.00 (116.28)
  Medium small LDL, change to last observation | 35.70 (52.40) | -11.47 (84.73)
  Small LDL, baseline | 878.68 (481.65) | 977.84 (622.99)
  Small LDL, change to last observation | 128.55 (236.89) | -74.09 (428.13)
  Very small LDL, baseline | 703.63 (385.31) | 780.78 (508.24)
  Very small LDL, change to last observation | 92.75 (193.00) | -62.50 (347.08)
  VLDL mean particle size, baseline | 51.21 (8.57) | 51.05 (11.83)
  VLDL mean particle size, change to last observ. | 4.09 (7.83) | 1.80 (9.21)
Statistical Analysis 1: Comparison: Olanzapine; HDL particles, total; Test type: Superiority or Other; p = 0.009, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 2: Comparison: Risperidone; HDL particles, total; Test type: Superiority or Other; p = 0.959, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 3: Comparison: Olanzapine vs Risperidone; HDL particles, total; Test type: Superiority or Other; p = 0.038, ANCOVA — Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline TReatment Pooled Investigator
Statistical Analysis 4: Comparison: Olanzapine; IDL; Test type: Superiority or Other; p = 0.013, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 5: Comparison: Risperidone; IDL; Test type: Superiority or Other; p = 0.928, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 6: Comparison: Olanzapine vs Risperidone; IDL; Test type: Superiority or Other; p = 0.049, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 7: Comparison: Olanzapine; Medium small LDL; Test type: Superiority or Other; p = 0.009, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 8: Comparison: Risperidone; Medium small LDL; Test type: Superiority or Other; p = 0.662, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 9: Comparison: Olanzapine vs Risperidone; Medium small LDL; Test type: Superiority or Other; p = 0.12, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 10: Comparison: Olanzapine; Small LDL; Test type: Superiority or Other; p = 0.099, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 11: Comparison: Risperidone; Small LDL; Test type: Superiority or Other; p = 0.304, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 12: Comparison: Olanzapine vs Risperidone; Small LDL; Test type: Superiority or Other; p = 0.024, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 13: Comparison: Olanzapine; Very small LDL; Test type: Superiority or Other; p = 0.176, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 14: Comparison: Risperidone; Very small LDL; Test type: Superiority or Other; p = 0.246, t-test, 2 sided; Withn group p-values are from t-tests on LSMean change
Statistical Analysis 15: Comparison: Olanzapine vs Risperidone; Very small LDL; Test type: Superiority or Other; p = 0.033, ANCOVA — Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator
Statistical Analysis 16: Comparison: Olanzapine; VLDL mean particle size; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 17: Comparison: Risperidone; VLDL mean particle size; Test type: Superiority or Other; p = 0.047, t-test, 2 sided; Within group p-values are from t-tests on LSMean change
Statistical Analysis 18: Comparison: Olanzapine vs Risperidone; VLDL mean particle size; Test type: Superiority or Other; p = 0.221, ANCOVA; Overall p-values are from Type 3 sums of squares ANCOVA, Model: Change=Baseline Treatment Pooled Investigator

ADVERSE EVENTS:
Arm/Group | Olanzapine | Risperidone
Serious Adverse Events (participants affected / at risk) | 2/68 | 5/62
Other Adverse Events (participants affected / at risk) | 42/68 | 43/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=68) | Risperidone (N=62)
Asthma (Immune system disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 1 (2)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=68) | Risperidone (N=62)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 5 (6)
Discomfort (General disorders) | 5 (5) | 2 (2)
Weight increased (Investigations) | 11 (11) | 4 (4)
Increased appetite (Metabolism and nutrition disorders) | 5 (5) | 7 (7)
Headache (Nervous system disorders) | 7 (9) | 8 (12)
Sedation (Nervous system disorders) | 7 (8) | 4 (5)
Anxiety (Psychiatric disorders) | 1 (1) | 6 (6)
Insomnia (Psychiatric disorders) | 4 (5) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days